CLINICAL TRIAL: NCT05279170
Title: Para Tracheal Compression to Prevent Gastric Insufflation During Positive Pressure Ventilation With Facemask in Children Under General Anaesthesia: an Efficiency Study
Brief Title: MAsk VEntilation With Paratracheal Pressure In Children. Para Tracheal Compression to Prevent Gastric Insufflation in Children
Acronym: MAVEPPIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020_74; 2021-A01535-36 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-02-24; First posted 2022-03-15 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Surgery; Anesthesia Intubation Complication
Keywords: Low Left Paratracheal esophagus Pressure; gastric insufflation; Echography; children; elective surgery; positive pressure ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children (Experimental): Compression of adjacent vessels (jugular vein and carotid artery), near the left paratracheal area. The risk of compression of the vessels will be assessed before performing the maneuver.
  At the screening time before the intervention, we will perfom an ultrasonography measurement while we applied the maneuver in order to eliminate a risk of compression of the vessels, defined as a reduction in diameter of 50%.
  Interventions: Other: MAVEPPIC: MAsk VEntilation with Paratracheal Pressure In Children

INTERVENTIONS:
Other: MAVEPPIC: MAsk VEntilation with Paratracheal Pressure In Children — Pressure will be applied with two fingers in the area located between the trachea and the sternal head of the sternocleidomastoid muscle on the left side to compress the cervical esophagus.
  The force applied (after measuring the equivalent force applied on a precision scale) will be about 10 - 15 N. This force will be adapted according to the child's body weight : 10 N below 20 kgs and 15 N between 20 kgs and 40 kgs

SUMMARY:
The use of cricoid pressure to prevent gastric aspiration or regurgitation in case of "full stomach" situation or emergency is still controversial in the adult population. Moreover this maneuver is no more recommended in children by some European pediatric anesthesia societies, because of a lack of evidence of its protective effect against gastric aspiration and its possible adverse effects.

A new approach to occlude effectively the esophageal lumen has been recently described in adults and has shown its effectiveness to prevent gastric insufflation. But this maneuver has so far not been evaluated in the pediatric population and could be an alternative to prevent gastro-esophageal regurgitation and pulmonary aspiration in children

ELIGIBILITY:
Inclusion Criteria:

* Children from 2 to 10 years of age who benefit from general anesthesia with or without intubation
* inhalation induction
* elective surgery
* ASA status 1 or 2
* consent of the child if he/she is able to express it
* consent of both parents and/or legal guardians
* socially insured

Exclusion Criteria:

* Child under 2 years old or > 10 years
* body weight is over 40 kgs
* ASA status 3 or higher
* Emergency surgery or unscheduled surgery
* scheduled ENT or esogastric surgery
* Achalasia of the esophagus or history of GERD pathology
* History of esophageal surgery (NISSEN type)
* BMI indexed to age and sex showing childhood obesity
* Predictable mask ventilation difficulties
* History of Tracheostomy
* Child not insured by social security

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Presence of air artefacts during positive pressure ventilation as evaluated by simultaneous gastric ultrasonography | We will perfom a unique measurement of gastric air artefact by ultrasonography after 2 minutes of positive pressure ventilation.
  Presence of antral and/or gastric air artefact described in ultrasonography. US will be perform during positive pressure mask ventilation.

SECONDARY OUTCOMES:
The verification of the actual position of the esophagus on the left side of the trachea at the place where LPPP will be applied (feasibility of LLPP) | Before the beginning of positive pressure ventilation during 1 minute
  Left side of the trachea ultrasonography performed before positive pressure ventilation
The safety of the LLPP maneuver: absence of any significant compression of the adjacent vessels as measured by US. | Before the beginning of positive pressure ventilation and during 1 minute
  Left side of the trachea ultrasonography performed before positive pressure ventilation
The expired tidal volume and peak inspiratory pressure as measured during PPV to evaluate any difficulty in mask ventilation induced by LLPP. | At the beginning of positive pressure ventilation and during two minutes
  Expired tidal volume measured exhaled flow on anesthesia ventilator

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Jeanne de Flandre - Pôle Anesthésie Réanimation Pédiatrique, Lille, France